CLINICAL TRIAL: NCT03971812
Title: Organoids Derived From Induced-Pluripotent Stem Cells (iPS) From Patients
Brief Title: Organoids Derived From Induced-Pluripotent Stem Cells (iPS) From Patients With High Grade Astrocytoma
Acronym: GLIOMANOID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01; 2019-A00145-52 (Other: ID RCB number); RCAPHM19_0001 (Other: AP-HM secondary number)
Record Dates: First submitted 2019-05-31; First posted 2019-06-03 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with high grade astrocytoma: Patients meeting inclusion and non-inclusion criteria and having signed informed consent will be included in the study
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — A blood sample of two 10 mL ethylenediaminetetraacetic (EDTA) tubes will be taken at the time of the visit. This sample will be centrifuged for isolation of peripheral blood mononuclear cells (PBMC).

SUMMARY:
The objective of this study research proposal is to model human gliomagenesis using 3-Dimensional (3D) brain organoids derived from human induced pluripotent stem cells (hiPSCs).

The working hypothesis is that 3D brain organoids can develop glioma-like structures and recapitulate phenotypic traits of gliomas when generated from hiPSCs expressing genetic mutants associated with glioma predisposition.

Methodology : To develop this pioneer study on the use of hiPSC-based brain organoids as a strategy to model gliomagenesis and study the impact of genetic mutants, it will be collect the peripheral blood mononuclear cell from 20 patients with high grade astrocytoma with or without IDH mutation. iPS will be generated from these PBMC and will be genetically modified according to different mutations. Then, it will be generate brain organoids according to standard protocols. Brain organoids generated from all different cells will be collected at different time points and analyzed for the presence of glioma-like structures and phenotypic hallmarks of gliomas.

From the proposed experiments, it will be expect that brain organoids will develop glioma-like features upon the presence of genetic mutations. Thus, it will be expect to demonstrate that brain organoids can be used as a reliable strategy to test the impact of genetic mutants, including the possible synergistic cooperation between different mutations on early gliomagenic events.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged 18 years or older
* Astrocytoma grades 3 or 4, confirmed by anatomopathological diagnosis
* Patient having signed an informed consent

Exclusion Criteria:

* Person in emergency situation, a legal person of legal age (guardianship, guardianship or legal guardianship), or unable to express his / her consent
* No affiliation to a social security scheme (beneficiary or beneficiary)
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients managed for a brain tumor for whom a blood sample collected routinely will be recovered
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-06-07 (Estimated); Primary Completion 2020-12-06 (Estimated); Study Completion 2020-12-06 (Estimated)

PRIMARY OUTCOMES:
Characterize the level of proliferation of organoids | 18 months
  compare different immunohistochemical markings between organoids

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No